CLINICAL TRIAL: NCT00980330
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Trial to Investigate the Efficacy, Tolerability, Safety and Pharmacokinetics of TMC435 as Part of a Treatment Regimen Including PegIFNa-2a and Ribavirin in HCV Genotype 1 Infected Subjects Who Failed Previous Standard Therapy
Brief Title: A Safety and Effectiveness Study of TMC435 in Chronic, Genotype 1, Hepatitis C Patients Who Failed to Previous Standard Treatment
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016063; TMC435-TiDP16-C206 (Other: Tibotec Pharmaceuticals, Ireland); 2009-010590-20 (EudraCT Number)
Record Dates: First submitted 2009-09-10; First posted 2009-09-21 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Peginterferon alpha-2a; PegIFNalpha-2a; RBV; Ribavirin; Placebo; TMC435-TIDP16-C206; TMC435-C206; TMC435; HCV
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- TMC435 100 mg 12 Wks + PR48 (Experimental): Participants will receive TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo with PR for 36 weeks.
  Interventions: Drug: TMC435; Drug: Placebo; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- TMC435 100 mg 24 Wks + PR48 (Experimental): Participants willl receive TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks followed by Placebo with PR for 24 weeks.
  Interventions: Drug: TMC435; Drug: Placebo; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- TMC435 100 mg 48 Wks + PR48 (Experimental): Participants will receive TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
  Interventions: Drug: TMC435; Drug: Placebo; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- TMC435 150 mg 12 Wks + PR48 (Experimental): Participants will receive TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo and PR for 36 weeks.
  Interventions: Drug: TMC435; Drug: Placebo; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- TMC435 150 mg 24 Wks + PR48 (Experimental): Participants will receive TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks followed Placebo and PR for 24 weeks.
  Interventions: Drug: TMC435; Drug: Placebo; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- TMC435 150 mg 48 Wks + PR48 (Experimental): Participants will receive TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
  Interventions: Drug: TMC435; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)
- Placebo 48 Wks + PR48 (Placebo Comparator): Participants will receive Placebo once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
  Interventions: Drug: TMC435; Drug: Peg-IFN-alfa-2a (P); Drug: Ribavirin (R)

INTERVENTIONS:
Drug: TMC435 — One TMC435 100-mg capsule or two 75-mg capsules orally (by mouth) once daily for 12, 24, or 48 weeks.
Drug: Placebo — One or 2 capsules of placebo identical in appearance to TMC435 taken orally once daily for 24, 36, or 48 weeks.
  Arms: TMC435 100 mg 12 Wks + PR48; TMC435 100 mg 24 Wks + PR48; TMC435 100 mg 48 Wks + PR48; TMC435 150 mg 12 Wks + PR48; TMC435 150 mg 24 Wks + PR48
Drug: Peg-IFN-alfa-2a (P) — 180 micrograms taken as one 0.5 mL subcutaneous injection once weekly for 48 weeks.
  Other Names: PEGASYS
Drug: Ribavirin (R) — 1000 or 1200 mg/day (5 or 6 tablets) taken orally as a twice daily regimen taken for 48 weeks.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of different regimens of TMC435 with standard treatment compared to standard treatment alone in participants with chronic, genotype 1, hepatitis C virus (HCV) infection who has failed previous treatment with pegylated interferon (Peg-INF-alfa-2a) and ribavirin (RBV).

DETAILED DESCRIPTION:
The study is a randomized (study drug assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled Phase IIb trial with TMC435 in participants with chronic, genotype 1, hepatitis C virus (HCV) infection who have failed standard treatment with pegylated interferon (Peg-INF-alfa-2a) and ribavirin (RBV). The study will compare the efficacy, tolerability and safety of different regimens with TMC435 combined with standard treatment (Peg-INF-alfa-2a and RBV) versus standard treatment alone. The trial will consist of a screening period of maximum 6 weeks, a 48-week treatment period, and a 24-week follow-up period. Participants will be eligible to enroll in the trial if they failed to respond to a prior course of standard treatment or relapsed following standard treatment. Participants will be randomly assigned to receive TMC435 with standard treatment for 12 weeks followed by standard treatment (plus placebo) for 36 weeks, TMC435 (100 mg or 150 mg once a day) with standard treatment for 24 weeks followed by standard treatment (plus placebo) for 24 weeks, TMC435 (100 mg or 150 mg once a day) with standard treatment for 48 weeks, or a placebo with standard treatment for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have chronic hepatitis C infection as evidenced by liver biopsy, anti-hepatitis C virus (HCV) and HCV RNA positive
* Must have chronic hepatitis C infection (genotype 1) with HCV RNA level greater than10000 IU/mL
* Patient must have failed at least 1 prior course of peg interferon (Peg-IFN-alfa-2a)/ribavirin (RBV) therapy (standard treatment)
* Must be willing to use 2 effective methods of birth control for up to 7 months after last dose of study medication

Exclusion Criteria:

* Has an evidence of decompensated liver disease
* Co-infection with any other Hepatitis C virus genotype or co-infection with the human immunodeficiency virus (HIV)
* Has a medical condition which is a contraindication to Peg-INF or RBV therapy
* Have had history of, or any current medical condition which could impact the safety of the patient in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (78):
- United States (17):
  - La Jolla, California
  - Los Angeles, California
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Laurel, Maryland
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Germantown, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
- Australia (8):
  - Concord
  - Darlinghurst
  - Fitzroy
  - Melbourne
  - New Lambton Heights
  - Parkville
  - Sydney
  - Woolloongabba
- Vienna, Austria
- Belgium (6):
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Roeselare
- Canada (4):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (6):
  - Créteil
  - Grenoble
  - Lyon
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (8):
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt A. M.
  - Freiburg im Breisgau
  - Hanover
  - Stuttgart
  - Würzburg
- Israel (7):
  - Haifa
  - Jerusalem
  - Nazareth
  - Petah Tikva
  - Ramat Gan
  - Safed
  - Tel Aviv
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- Norway (3):
  - Nordbyhagen
  - Oslo
  - Tromsø
- Poland (5):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Kielce
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (5):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Smolensk
- United Kingdom (2):
  - London
  - Plymouth

REFERENCES:
- [Derived] Lenz O, Verbinnen T, Fevery B, Tambuyzer L, Vijgen L, Peeters M, Buelens A, Ceulemans H, Beumont M, Picchio G, De Meyer S. Virology analyses of HCV isolates from genotype 1-infected patients treated with simeprevir plus peginterferon/ribavirin in Phase IIb/III studies. J Hepatol. 2015 May;62(5):1008-14. doi: 10.1016/j.jhep.2014.11.032. Epub 2014 Nov 28. PMID 25445400
- [Derived] Scott J, Rosa K, Fu M, Cerri K, Peeters M, Beumont M, Zeuzem S, Evon DM, Gilles L. Fatigue during treatment for hepatitis C virus: results of self-reported fatigue severity in two Phase IIb studies of simeprevir treatment in patients with hepatitis C virus genotype 1 infection. BMC Infect Dis. 2014 Aug 26;14:465. doi: 10.1186/1471-2334-14-465. PMID 25164700
- [Derived] Zeuzem S, Berg T, Gane E, Ferenci P, Foster GR, Fried MW, Hezode C, Hirschfield GM, Jacobson I, Nikitin I, Pockros PJ, Poordad F, Scott J, Lenz O, Peeters M, Sekar V, De Smedt G, Sinha R, Beumont-Mauviel M. Simeprevir increases rate of sustained virologic response among treatment-experienced patients with HCV genotype-1 infection: a phase IIb trial. Gastroenterology. 2014 Feb;146(2):430-41.e6. doi: 10.1053/j.gastro.2013.10.058. Epub 2013 Nov 1. PMID 24184810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 89 sites in 14 countries.
Pre-assignment Details: A total of 618 participants were screened. Of these, 463 participants were randomized of whom 462 participants started treatment. One participant in the placebo group was 'randomized in error,' did not receive treatment, and was withdrawn from the study due to non-compliance (did not come for visit).
Groups:
- TMC435 100mg 12 Wks + PR48: Participants received TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo with PR for 36 weeks.
- TMC435 100mg 24 Wks + PR48: Participants received TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks followed by Placebo with PR for 24 weeks.
- TMC435 100mg 48 Wks + PR48: Participants received TMC435 100 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
- TMC435 150mg 12 Wks + PR48: Participants received TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 12 weeks followed by Placebo and PR for 36 weeks.
- TMC435 150mg 24 Wks + PR48: Participants received TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 24 weeks followed Placebo and PR for 24 weeks.
- TMC435 150mg 48 Wks + PR48: Participants received TMC435 150 mg once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
- Placebo 48Wks + PR48: Participants received Placebo once daily with Peg-IFN-alfa-2a (P) once weekly and ribavirin (R) twice daily for 48 weeks.
Period: Overall Study
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Started | 66 | 65 | 66 | 66 | 68 | 65 | 66
Completed | 61 | 60 | 58 | 61 | 63 | 61 | 59
Not Completed | 5 | 5 | 8 | 5 | 5 | 4 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 4 | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 1 | 3 | 2 | 5
Not completed — (not specified) | 2 | 0 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48 | Total
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66 | 462
Age, Continuous [Median (Full Range); unit: years] | 51.5 [20 to 68] | 50 [20 to 68] | 50 [22 to 69] | 48 [20 to 63] | 51.5 [25 to 68] | 50 [21 to 69] | 50.5 [22 to 66] | 50 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 21 | 21 | 25 | 17 | 24 | 151
  Male | 44 | 44 | 45 | 45 | 43 | 48 | 42 | 311
Region of Enrollment [Number; unit: participants]
  Asia Pacific | 4 | 5 | 4 | 4 | 1 | 4 | 7 | 29
  Europe and Israel | 34 | 46 | 46 | 49 | 49 | 43 | 46 | 313
  North-America | 28 | 14 | 16 | 13 | 18 | 18 | 13 | 120
Prior PR response [Number; unit: participants] — In the study, "Null Responders" were participants with less than 2 log10 IU/mL reduction in HCV RNA compared to baseline at Week 12 of the previous PegIFNα-2a/b and RBV treatment; "Partial Responders" were participants with a greater than or equal to 2 log10 IU/mL reduction in HCV RNA compared to baseline at Week 12, but not achieving an undetectable HCV RNA at the end of the previous PegIFNα-2a/b and RBV treatment; and "Relapsers" were participants with HCV RNA undetectable at end of the previous treatment with PegIFNα-2a/b and RBV, but detectable HCV RNA within 24 weeks of follow-up.
  participants
    Null responder | 16 | 16 | 18 | 17 | 17 | 17 | 16 | 117
    Partial responder | 23 | 23 | 22 | 23 | 24 | 22 | 23 | 160
    Relapser | 27 | 26 | 26 | 26 | 27 | 26 | 27 | 185
Metavir Score [Number; unit: participants] — A Metavir score is used to interpret the degree of inflammation and fibrosis in a liver biopsy. Below are fibrosis scores graded on a 5-point scale from F0 (no fibrosis) to F4 (cirrhosis).
  participants
    Not reported | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 7
    Score F0 | 6 | 3 | 6 | 5 | 11 | 1 | 7 | 39
    Score F1 | 17 | 14 | 23 | 19 | 11 | 27 | 18 | 129
    Score F2 | 21 | 17 | 9 | 18 | 21 | 16 | 16 | 118
    Score F3 | 14 | 16 | 14 | 11 | 11 | 7 | 13 | 86
    Score F4 | 7 | 13 | 14 | 13 | 13 | 13 | 10 | 83

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response at the End of Treatment (EOT) and 24 Weeks After the EOT (SVR24)
Description: The table below shows the percentage of participants in the overall population with an SVR24, defined as having plasma levels of Hepatitis C Virus ribonucleic acid less than 25 IU/mL undetectable at the EOT and 24 weeks after the EOT.
Time Frame: Week 72
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 69.7 | 66.2 | 60.6 | 66.7 | 72.1 | 80.0 | 22.7

2. Secondary Outcome: The Percentage of Participants With a Greater Than 2 log10 Drop in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at Time Points During Treatment
Description: The table below shows the percentage of participants in each treatment group who achieved a greater than 2 log10 drop in plasma levels of HCV RNA at selected time points during treatment.
Time Frame: Weeks, 2, 4, 8, and 12
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants
  Week 2 | 97.0 | 93.8 | 97.0 | 100.0 | 95.6 | 96.9 | 24.2
  Week 4 | 92.4 | 93.8 | 92.4 | 97.0 | 91.2 | 96.9 | 36.4
  Week 8 | 92.4 | 89.2 | 89.4 | 93.9 | 91.2 | 95.4 | 57.6
  Week 12 | 90.9 | 87.7 | 84.8 | 92.4 | 91.2 | 92.3 | 60.6

3. Secondary Outcome: The Percentage of Participants Achieving Plasma Levels of Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment who achieved plasma HCV RNA levels of <25 IU/mL undetectable at selected time points during treatment and follow-up and at the end of treatment (EOT).
Time Frame: Weeks, 2, 4, 8, 12, 24, 36, 48, 60, 72 and EOT (up to Week 48)
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants
  Week 2 | 22.7 | 18.5 | 15.2 | 24.2 | 32.4 | 27.7 | 0.0
  Week 4 | 66.7 | 58.5 | 53.0 | 62.1 | 67.6 | 66.2 | 1.5
  Week 8 | 77.3 | 75.4 | 77.3 | 84.8 | 83.8 | 83.1 | 7.6
  Week 12 | 81.8 | 73.8 | 72.7 | 80.3 | 85.3 | 83.1 | 19.7
  Week 24 | 81.8 | 75.4 | 78.8 | 83.3 | 86.8 | 86.2 | 42.4
  Week 36 | 78.8 | 73.8 | 78.8 | 80.3 | 83.8 | 81.5 | 39.4
  Week 48 | 81.8 | 73.8 | 74.2 | 75.8 | 80.9 | 81.5 | 37.9
  Week 60 | 69.7 | 67.7 | 59.1 | 66.7 | 72.1 | 76.9 | 22.7
  Week 72 | 69.7 | 66.2 | 60.6 | 66.7 | 73.5 | 80.0 | 22.7
  EOT (up to Week 48) | 80.3 | 78.5 | 80.3 | 80.3 | 83.8 | 86.2 | 40.9

4. Secondary Outcome: The Percentage of Participants Achieving Plasma Levels of Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Detectable or Undetectable During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment group who achieved plasma HCV RNA levels below the limit of quantification defined as less than 25 IU/mL (detectable or undetectable) at selected time points during treatment, follow-up, and at the end of treatment (EOT).
Time Frame: Weeks, 2, 4, 8, 12, 24, 36, 48, 60, 72, and EOT (up to Week 48)
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of Participants
  Week 2 | 60.6 | 55.4 | 54.5 | 63.6 | 60.3 | 66.2 | 3.0
  Week 4 | 78.8 | 72.3 | 81.8 | 86.4 | 82.4 | 86.2 | 3.0
  Week 8 | 87.9 | 81.5 | 84.8 | 87.9 | 89.7 | 87.7 | 12.1
  Week 12 | 87.9 | 81.5 | 83.3 | 89.4 | 88.2 | 89.2 | 34.8
  Week 24 | 84.8 | 78.5 | 80.3 | 86.4 | 86.8 | 89.2 | 50.0
  Week 36 | 81.8 | 73.8 | 78.8 | 81.8 | 86.8 | 84.6 | 43.9
  Week 48 | 83.3 | 73.8 | 74.2 | 78.8 | 82.4 | 81.5 | 40.9
  Week 60 | 71.2 | 67.7 | 60.6 | 66.7 | 72.1 | 78.5 | 22.7
  Week 72 | 69.7 | 66.2 | 60.6 | 66.7 | 73.5 | 80.0 | 22.7
  EOT (up to Week 48) | 86.4 | 81.5 | 81.8 | 89.4 | 89.7 | 89.2 | 47.0

5. Secondary Outcome: The Percentage of Participants Achieving a Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants in each treatment group who achieved a RVR, defined as having an undetectable plasma Hepatitis C virus ribonucleic acid level after receiving 4 weeks of treatment.
Time Frame: Week 4
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 66.7 | 58.5 | 53.0 | 62.1 | 67.6 | 66.2 | 1.5

6. Secondary Outcome: The Percentage of Participants Achieving an Early Virologic Response (EVR)
Description: The table below shows the percentage of participants who achieved an EVR, defined as having a greater than or equal to 2 log10 reduction in plasma Hepatitis C virus ribonucleic acid from baseline at Week 12.
Time Frame: Week 12
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 90.9 | 87.7 | 84.8 | 92.4 | 91.2 | 92.3 | 60.6

7. Secondary Outcome: The Percentage of Participants Achieving a Complete Early Virologic Response (cEVR)
Description: The table below shows the percentage of participants in each treatment group who had a cEVR, defined as having undetectable plasma levels of Hepatitis C virus ribonucleic acid at Week 12.
Time Frame: Week 12
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 81.8 | 73.8 | 72.7 | 80.3 | 85.3 | 83.1 | 19.7

8. Secondary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: The table below shows the percentage of participants in the overall population who achieved undetectable plasma Hepatitis C virus ribonucleic acid levels at the end of treatment (EOT) and 12 Weeks after the planned EOT.
Time Frame: Week 60
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 69.7 | 67.7 | 60.6 | 66.7 | 72.1 | 80.0 | 22.7

9. Secondary Outcome: The Percentage of Participants With Viral Breakthrough
Description: The table below shows the percentage of participants in the overall population in each treatment group during the treatment period who experienced viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in Hepatitis C virus (HCV) ribonucleic acid (RNA) from the lowest level reached or a confirmed HCV RNA of > 100 IU/mL in participants whose HCV RNA had previously been below the lower limit of quantification (i.e., less than 25 IU/mL detectable or undetectable).
Time Frame: EOT (up to Week 48)
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 10.6 | 13.8 | 13.6 | 9.1 | 10.3 | 7.7 | 1.5

10. Secondary Outcome: The Percentage of Participants With Viral Relapse
Description: The table below shows the percentage of participants in the overall population who had viral relapse, defined as confirmed detectable Hepatitis C virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with HCV RNA less than 25 IU/mL undetectable at end of treatment.
Time Frame: Up to Week 72
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Number analyzed (Participants) | 66 | 65 | 66 | 66 | 68 | 65 | 66
Percentage of participants | 9.3 | 13.7 | 18.0 | 11.8 | 14.0 | 5.5 | 44.4

11. Secondary Outcome: The Number of Participants Who Achieved Normalized Alanine Aminotransferase (ALT) Levels at the End of Treatment (EOT)
Description: The table below shows the number of participants with abnormal ALT levels at Baseline who achieved the normal ALT levels at the EOT (up to Week 48).
Time Frame: EOT (up to Week 48)
Population: Intent-to-treat: Participants who received at least 1 dose of study medication were included.
Measure: Number; unit: Percentage of participants
Groups:
- All TMC435: Participants in all 6 TMC435 treatment groups combined.
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | All TMC435
Number analyzed (Participants) | 36 | 49 | 45 | 40 | 43 | 43 | 256
Percentage of participants | 26 | 37 | 31 | 23 | 31 | 33 | 181

12. Secondary Outcome: Plasma Concentrations of TMC435
Description: The table below shows median (range) predose plasma concentration (C0h) values and median (range) average steady-state plasma concentration (Css,av) values for TMC435 for participants in each of the 6 TMC435 treatment groups.
Time Frame: 0 (predose, baseline) and 4, 8, 12, and 24 hours post-dose at Weeks 2, 4, 8, 12, 16, 24, and 48
Population: Participants who received at least 1 dose of study medication with at least 1 post-baseline pharmacokinetic (PK) assessment were included in the PK analysis population.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48
Number analyzed (Participants) | 66 | 65 | 65 | 66 | 68 | 64
ng/mL
  C0h | 380.5 [34 to 3599] | 411.3 [101 to 6943] | 529.8 [62 to 4212] | 1323.5 [37 to 12478] | 1074.0 [110 to 14303] | 886.1 [150 to 21825]
  Css,av | 691.1 [204 to 3960] | 770.5 [344 to 7218] | 892.0 [290 to 4580] | 1960.9 [304 to 13047] | 1792.3 [532 to 14892] | 1606.9 [635 to 22417]

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24h) for TMC435
Description: The table below shows the median (range) AUC24h values for TMC435 for participants in each TMC435 treatment group.
Time Frame: 0 (predose, baseline) and 4, 8, 12, and 24 hours post-dose at Weeks 2, 4, 8, 12, 16, 24, and 48
Population: as for outcome 12
Measure: Median (Full Range); unit: ng.h/mL
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48
Number analyzed (Participants) | 66 | 65 | 65 | 66 | 68 | 64
ng.h/mL | 16587.0 [4897 to 95030] | 18492.5 [8252 to 173240] | 21409.0 [6949 to 109920] | 47061.8 [7301 to 313135] | 43015.0 [12777 to 357415] | 38564.5 [15233 to 538010]

ADVERSE EVENTS:
Time Frame: Week 72
Arm/Group | TMC435 100mg 12 Wks + PR48 | TMC435 100mg 24 Wks + PR48 | TMC435 100mg 48 Wks + PR48 | TMC435 150mg 12 Wks + PR48 | TMC435 150mg 24 Wks + PR48 | TMC435 150mg 48 Wks + PR48 | Placebo 48Wks + PR48
Serious Adverse Events (participants affected / at risk) | 3/66 | 5/65 | 3/66 | 7/66 | 5/68 | 8/65 | 4/66
Other Adverse Events (participants affected / at risk) | 63/66 | 61/65 | 65/66 | 63/66 | 65/68 | 63/65 | 63/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100mg 12 Wks + PR48 (N=66) | TMC435 100mg 24 Wks + PR48 (N=65) | TMC435 100mg 48 Wks + PR48 (N=66) | TMC435 150mg 12 Wks + PR48 (N=66) | TMC435 150mg 24 Wks + PR48 (N=68) | TMC435 150mg 48 Wks + PR48 (N=65) | Placebo 48Wks + PR48 (N=66)
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia bordetella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100mg 12 Wks + PR48 (N=66) | TMC435 100mg 24 Wks + PR48 (N=65) | TMC435 100mg 48 Wks + PR48 (N=66) | TMC435 150mg 12 Wks + PR48 (N=66) | TMC435 150mg 24 Wks + PR48 (N=68) | TMC435 150mg 48 Wks + PR48 (N=65) | Placebo 48Wks + PR48 (N=66)
Fatigue (General disorders) | 30 | 28 | 34 | 26 | 28 | 28 | 29
Influenza like illness (General disorders) | 23 | 24 | 21 | 16 | 18 | 14 | 13
Asthenia (General disorders) | 6 | 16 | 11 | 16 | 16 | 19 | 7
Pyrexia (General disorders) | 6 | 10 | 13 | 14 | 17 | 9 | 9
Irritability (General disorders) | 9 | 8 | 10 | 8 | 10 | 8 | 7
Chills (General disorders) | 7 | 4 | 4 | 6 | 6 | 7 | 6
Injection site erythema (General disorders) | 3 | 4 | 1 | 3 | 3 | 7 | 2
Injection site reaction (General disorders) | 3 | 2 | 4 | 2 | 3 | 1 | 0
Pain (General disorders) | 1 | 2 | 1 | 4 | 2 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 26 | 21 | 20 | 25 | 24 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 15 | 12 | 14 | 10 | 12 | 10
Rash (Skin and subcutaneous tissue disorders) | 8 | 8 | 6 | 10 | 13 | 16 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3 | 7 | 7 | 6 | 7 | 5
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5 | 7 | 3 | 5 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 5 | 3 | 0 | 1 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 3 | 7 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 1 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 17 | 10 | 20 | 20 | 11 | 17 | 14
Diarrhoea (Gastrointestinal disorders) | 9 | 11 | 13 | 9 | 8 | 9 | 13
Dry mouth (Gastrointestinal disorders) | 6 | 4 | 4 | 3 | 4 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 1 | 2 | 6 | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2 | 5 | 6 | 3 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 4 | 5 | 4 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 4 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 3 | 4 | 0
Toothache (Gastrointestinal disorders) | 1 | 4 | 2 | 2 | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 4 | 2 | 0 | 0 | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 18 | 19 | 23 | 29 | 26 | 23 | 24
Dizziness (Nervous system disorders) | 1 | 4 | 7 | 6 | 4 | 7 | 6
Disturbance in attention (Nervous system disorders) | 3 | 8 | 5 | 1 | 3 | 5 | 3
Dysgeusia (Nervous system disorders) | 5 | 2 | 6 | 6 | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 11 | 11 | 16 | 11 | 20 | 10 | 9
Depression (Psychiatric disorders) | 7 | 8 | 8 | 10 | 6 | 6 | 6
Sleep disorder (Psychiatric disorders) | 5 | 2 | 5 | 7 | 2 | 5 | 2
Anxiety (Psychiatric disorders) | 5 | 2 | 3 | 2 | 2 | 3 | 3
Depressed mood (Psychiatric disorders) | 2 | 2 | 3 | 0 | 2 | 5 | 3
Mood altered (Psychiatric disorders) | 2 | 0 | 3 | 4 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 16 | 15 | 15 | 17 | 18 | 20 | 11
Anaemia (Blood and lymphatic system disorders) | 14 | 11 | 12 | 10 | 16 | 13 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 7 | 6 | 5 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 4 | 3 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 13 | 11 | 8 | 16 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 8 | 4 | 8 | 10 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4 | 2 | 3 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 4 | 2 | 1 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1 | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 3 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 4 | 6 | 11 | 11 | 16 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 9 | 15 | 7 | 7 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 3 | 9 | 2 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 3 | 4 | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 7 | 1 | 2 | 4 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 3 | 3 | 4 | 1 | 5
Sinusitis (Infections and infestations) | 7 | 0 | 3 | 1 | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 2 | 0 | 3 | 2
Weight decreased (Investigations) | 4 | 3 | 3 | 5 | 3 | 7 | 3
Neutrophil count decreased (Investigations) | 2 | 5 | 0 | 2 | 1 | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 1 | 0 | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 3 | 4 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 11 | 11 | 13 | 13 | 10 | 9
Dry eye (Eye disorders) | 1 | 4 | 4 | 0 | 3 | 2 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2 | 0 | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 1 | 2 | 2 | 7 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 4 | 0 | 3 | 1 | 4
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 0 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days